CLINICAL TRIAL: NCT05363540
Title: Optimal Timing of Parasternal Intercostal Nerve Block Application (Pre-incisional Versus Post-incisional) for Acute Pain Management in Cardiac Surgery; a Randomized Double Blinded Clinical Trial
Brief Title: Optimal Timing of Parasternal Intercostal Nerve Block Application for Acute Pain Management in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Samar Rafik Mohamed Amin, lecturer of anesthesia and surgical ICU, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RC.1-3-2022
Record Dates: First submitted 2022-04-17; First posted 2022-05-06 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Pain, Acute
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-incisional parasternal block (Active Comparator): ultrasound guided parasternal intercostal block will be administrated before surgical incision.
  Interventions: Procedure: pre-incisional parasternal intercostal block
- Post-incisional parasternal block (Active Comparator): under direct vision parasternal intercostal block will be administrated after surgical incision and before closure of the sternum.
  Interventions: Procedure: post-incisional parasternal intercostal block

INTERVENTIONS:
Procedure: pre-incisional parasternal intercostal block — LA will be administrated by the anesthesiologist under ultrasound guidance and before surgical incision On either side of thorax, 2 cm lateral to sternal edge from 2nd to 6th intercostal space, A volume of (4 mL) of 0.25% bupivacaine will be used
  Arms: Pre-incisional parasternal block
Procedure: post-incisional parasternal intercostal block — LA will be administered by the cardiac surgeon before the sternal closure. injection will introduced 2 cm lateral to sternal edge from 2nd to 6th intercostal space and volume (4 mL) of 0.25% bupivacaine will be used.
  Arms: Post-incisional parasternal block

SUMMARY:
Patients experiencing pain after undergoing cardiac surgery may also experience prolonged immobilization, insufficient respiratory functions, and the inability to cough due to median sternotomy. Therefore, duration of mechanical ventilation, length of intensive care unit (ICU) stay, and length of hospital stay of these patients will increase significantly.

many facial plane blocks have been introduced as simple and safe intervention for thoracic wall anesthesia and analgesia. Parasternal intercostal nerve block (PSIB) is a "superficial block" which involves local anesthetic (LA) infiltration in the intercostal space around the sternum where the anterior branches of intercostal nerves exist.

Intraoperative LA administration under direct vision of the surgeon ensures adequate delivery of drugs and minimizes bleeding complication or inadvertent administration in blood vessels. Meanwhile, Preoperative administration of LA guided by ultrasound imaging has been used in variable surgical settings with noticeable success because of preemptive inhibition of noxious stimuli.

ELIGIBILITY:
Inclusion Criteria:

* Age from 20-70 years,
* Scheduled to undergo elective cardiac surgeries through median sternotomy involving cardiopulmonary bypass (CPB).

Exclusion Criteria:

* Patients requiring preoperative inotropes, mechanical ventilation or intra-aortic balloon pump,
* patients who have previous cardiac surgery,
* prolonged CPB time (CPB>120 minutes),
* Intubation time more than 12hrs or planned for overnight ventilation.
* Allergy to any of used drugs,
* opioids addiction,
* Chronic liver disease, chronic renal disease, and cognitive impairment.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2022-12-24 (Actual)

PRIMARY OUTCOMES:
Amount of rescue analgesia | 24 hours postoperative
  Total amount of opioid administered as rescue analgesia postoperative.

SECONDARY OUTCOMES:
Intraoperative total fentanyl requirements | during surgery
  the amount of consumed opioid during the procedure
intraoperative mean arterial blood pressure (MAP) | during surgery (baseline, at skin incision, at sternotomy, at sternal retraction)
  hemodynamic variability due to surgical stimulation
pain score (VAS) | at extubation, 12th, 16th, 20th, and 24th hour postoperative
  VAS scores will be recorded by making a handwritten mark on a 10-cm line that represented a continuum between "no pain" and "worst possible pain."
adverse effects | 24 hours postoperative
  nausea, vomiting, excessive sedation, respiratory depression
patient satisfaction | 28 hours postoperative
  0 "extremely unsatisfied" to 10 "extremely satisfied"
Intensive Care Unit (ICU) Length of Stay | up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Samar Rafik Amin, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided